CLINICAL TRIAL: NCT03964116
Title: Impact of Sick Peer Relation on the Adaptation to Disease and on Treatment of Cancer-suffering Adolescents and Young Adults (PEERS-AYA)
Brief Title: Impact of Sick Peer Relation on Adaptation to Disease and on Treatment of Cancer-suffering Adolescents & Young Adults
Acronym: PAIRS-AJA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC 2017-10
Record Dates: First submitted 2018-11-02; First posted 2019-05-28 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Adolescent Behavior; Young Adult
MeSH Terms: conditions — Neoplasms; Adolescent Behavior | interventions — Interview, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AYA (Other): Questionnaires set all 3 months and psychological interviews if needed
  Interventions: Other: Questionnaires set all 3 months

INTERVENTIONS:
Other: Questionnaires set all 3 months — This longitudinal study based upon repeated and multicentric measurement will recruit AYA with cancer in care Units dedicated to them or not. Measures will be quantitative, and repeated every 3 months by questionnaires, as well as qualitative (social network questionnaire, psychological research interview) for teenagers declaring a negative event or a death event during treatments.
  Those patients presenting a high depression score will be contacted by a research psychologist for semi-directed interview.
  Other Names: Psychological interviews

SUMMARY:
Adolescents and young adults (AYA) with cancer have to deal with a relatively segmented organization of care between pediatric and adult medicine structures in France. However, the third french Plan Cancer 2014-2019 helped in the recognition of the specificities of the AYA affected by cancer and allowed the creation of specific structures in some care units in France, whose primary goal is the preservation of the social link.

Indeed, peer relations contribute to access to quality social support, which is an important variable in patient adjustment with cancer. The adolescents that perceive higher social support report less psychological distress and exhibit higher adaptation scores.

It nevertheless happens that AYA experience negative social support, often from friends because of contact reduction during the disease. Patients can then elect to turn towards non-intimate relations such as support groups. The main risk when a AYA with cancer defines a sick peer as one bringing him quality social support is the installation of a sense of guilt, for example, when a young person is confronted with disease negative progress or with peer death. The more an adolescent identifies with the deceased, the more he is able to consider his own mortality.

AYA units are developing in France, creating a community of sick adolescents. These communities are precious for AYA and allow information and experience sharing, a feeling of reduced isolation and a greater emotional closeness with peers suffering from the same disease.

How is social support from peers and close friends perceived by these young people in AYA units and through the social networks? What can the consequences of the evolution of peer disease be on AYA? What is the impact of the mourning of sick peers on these young people? What are the predictors?

DETAILED DESCRIPTION:
Methodology: Multicentric, prospective, not randomized study.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents or young adults from 15 to 27 years old (included) receiving cancer diagnose or recurrence announcement.
2. Patient information and free consent signature by the patient or his legal representative(s).

Exclusion Criteria:

1. Patient with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol.
2. Inability to understand, talk or write in French.
3. Patient individually deprived of liberty or placed under the authority of a tutor.

Ages: 15 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Social support on patients psychological adjustment | 4 years
  Compare the social support received and its effects on psychological adjustment in AYA unit groups versus groups without AYA unit (socio-demographic questionnaire).
Social support on patients psychological adjustment | 4 years
  Compare the social support received and its effects on psychological adjustment in AYA unit groups versus groups without AYA unit (BDI-II questionnaire).
Social support on patients psychological adjustment | 4 years
  Compare the social support received and its effects on psychological adjustment in AYA unit groups versus groups without AYA unit (STAI-Y questionnaire).
Psychological adjustment & quality | 4 years
  Compare psychological adjustment in the 2 groups and its quality according to important events (positive or negative) that affect sick peers (STAI-Y questionnaire).
Psychological adjustment & quality | 4 years
  Compare psychological adjustment in the 2 groups and its quality according to important events (positive or negative) that affect sick peers (BDI-II questionnaire).
Predictors of the grief quality | 4 years
  Define if there are predictors of the grief quality: personality? Attachment? Other life events? Depression? Nature of the link with dead peers? (RSQ questionnaire).
Predictors of the grief quality | 4 years
  Define if there are predictors of the grief quality: personality? Attachment? Other life events? Depression? Nature of the link with dead peers? (SSQ6 questionnaire).
Predictors of the grief quality | 4 years
  Define if there are predictors of the grief quality: personality? Attachment? Other life events? Depression? Nature of the link with dead peers? (BFI-Fr questionnaire).
Grief phenomenon (real or virtual life) | 4 years
  Describe the grief phenomenon and observe if there are demonstrations of grief when the peer was never met in person (ITG questionnaire).
Grief phenomenon (real or virtual life) | 4 years
  Describe the grief phenomenon and observe if there are demonstrations of grief when the peer was never met in person (SEC questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Valérie LAURENCE, MD, Principal Investigator — Institut Curie Paris; Cécile FLAHAULT, PhD, Study Director — Université René Descartes, Paris
Locations (2):
- France (2):
  - Centre Leon Berard, Lyon
  - INSTITUT CURIE - site Paris, Paris, Île-de-France Region

REFERENCES:
- [Background] Phan J, Vander Haegen M, Karsenti L, Laurence V, Marec-Berard P, Cordero C, Thisse A, Riberon C, Flahault C. Psychological Adjustment, Adaptation, and Perception of Social Support in French Adolescents and Young Adults After the Diagnosis of Cancer. J Adolesc Young Adult Oncol. 2023 Jun;12(3):389-397. doi: 10.1089/jayao.2022.0034. Epub 2022 Sep 6. PMID 36067271
- [Result] Phan J, Laurence V, Marec-Berard P, Cordero C, Riberon C, Flahault C. The Place of Sick Peers in Adolescents and Young Adults with Cancer: Advantage, Disadvantage, and What Makes Barriers to the Encounter. J Adolesc Young Adult Oncol. 2023 Dec;12(6):879-889. doi: 10.1089/jayao.2022.0176. Epub 2023 Mar 30. PMID 36999900